CLINICAL TRIAL: NCT01098929
Title: Gene Mutations and Rescue in Human Congenital Diaphragmatic Hernia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Patricia Donahoe, MD, Principal Investigator and Program Director, Pediatric Surgical Research Laboratories, Massachusetts General Hospital
Other Study IDs: 05-07-105R
Record Dates: First submitted 2010-03-31; First posted 2010-04-05 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: genes; genetic; chromosome; chromosome microarray
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, tissue, saliva, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Congenital Diaphragmatic Hernia (CDH): Individuals affected with congenital diaphragmatic hernia (CDH)
- Unaffected: Healthy family members of individuals affected with congenital diaphragmatic hernia (CDH)

SUMMARY:
Congenital diaphragmatic hernia (CDH) occurs when the diaphragm, the muscle that separates the chest cavity from the abdominal cavity, does not form properly. When an opening is present in the diaphragm, organs that are normally found in the abdomen can move up into the chest cavity. The primary objective of this study is to generate information about the hereditary basis of congenital diaphragmatic hernia and abnormal lung development. Our long-term goal is to identify ways to treat babies in utero with effective but safe drugs to speed up lung development before birth.

DETAILED DESCRIPTION:
This study uses a combination of clinical, molecular biological, and developmental strategies to better understand the genetic basis of congenital diaphragmatic hernia. Ongoing projects at Massachusetts General Hospital include identification of novel genes affecting diaphragm and lung development in a) mouse models using laser capture, microdissection, expression arrays, and statistical and bioinformatics analysis and b) human kindreds with multiple affected family members using linkage analysis and exome sequencing.

Research projects based at Children's Hospital Boston include a) continued recruitment of a population of patients with congenital diaphragmatic hernia who are carefully phenotyped for entry into an extensive database, b) collection of biological samples belonging to the phenotyped cohort of patients, c) next-generation sequencing on candidate genes and d) molecular cytogenetic studies such as comparative genomic hybridization and subtelomeric fluorescence in situ hybridization.

Over 500 patients with congenital diaphragmatic hernia and their families have been recruited to date and efforts are ongoing to double this number. The investigators hope that the information gained through identifying the genes that contribute to congenital diaphragmatic hernia will provide the foundation for future efforts to develop effective interventions for the treatment of this disease.

ELIGIBILITY:
Inclusion Criteria:

All individuals affected with a congenital diaphragmatic hernia (CDH), or with a family history of CDH

Exclusion Criteria:

Individuals with no personal or family history of a CDH

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children/infants with a congenital diaphragmatic hernia
  Women who are currently pregnant with a fetus diagnosed with congenital diaphragmatic hernia
  Individuals with a family history of congenital diaphragmatic hernia
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2002-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
identify genes associated with CDH | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Donahoe, MD, Principal Investigator — Massachusetts General Hospital; Jay Wilson, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States